CLINICAL TRIAL: NCT05998408
Title: A Phase I/II Study of the JAK1/2 Inhibitor Ruxolitinib for Relapsed / Refractory Immune Bone Marrow Failure
Brief Title: JAK1/2 Inhibitor Ruxolitinib for Relapsed/Refractory Immune Bone Marrow Failure
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10001667; 001667-H
Record Dates: First submitted 2023-08-17; First posted 2023-08-21 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12-17

CONDITIONS: Severe Aplastic Anemia; Single Lineage Cytopenias, T-LGL; Hypoplastic MDS
Keywords: Hematologic toxicity; Ruxolitinib
MeSH Terms: conditions — Anemia, Aplastic | interventions — ruxolitinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Subjects with hypoplastic MDS (Experimental): Subjects are defined as patients with a diagnosis of hMDS clinically confirmed by a licensed physician or an advanced practitioner who meets the inclusion and exclusion criteria and can provide informed consent.
  Interventions: Drug: Ruxolitinib
- Subjects with MAA (Experimental): Subjects are defined as patients with a diagnosis of MAA clinically confirmed by a licensed physician or an advanced practitioner who meets the inclusion andexclusion criteria and can provide informed consent.
  Interventions: Drug: Ruxolitinib
- Subjects with PRCA (Experimental): Subjects are defined as patients with a diagnosis of PRCA clinically confirmed by a licensed physician or advanced practitioners who meet the inclusion and exclusion criteria and can provide informed consent.
  Interventions: Drug: Ruxolitinib
- Subjects with SAA (Experimental): Subjects are defined as patients with a diagnosis of SAA clinically confirmed by a licensed physician oran advanced practitioner who meets the inclusion andexclusion criteria and can provide informed consent.
  Interventions: Drug: Ruxolitinib
- Subjects with TLGL (Experimental): Subjects are defined as patients with a diagnosis of TLGL clinically confirmed by a licensed physician or advanced practitioner who meets the inclusion and exclusion criteria and can provide informed consent.
  Interventions: Drug: Ruxolitinib

INTERVENTIONS:
Drug: Ruxolitinib — Subjects will be instructed to take ruxolitinib at up to 20mg (total) BID for up to 6 months (with or without food)

SUMMARY:
Background:

Immune bone marrow failure is a condition that occurs when a person s immune system attacks the cells of the bone marrow. This can lead to diseases including different types of anemias and blood cancers. Some of these diseases can be deadly. Better treatments are needed.

Objective:

To test a drug (ruxolitinib) in people with different types of immune bone marrow failure.

Eligibility:

Adults aged 18 and older with an immune bone marrow failure.

Design:

Participants will be screened. They will have a physical exam. They will give samples of blood and saliva. They will have a bone marrow biopsy: A large needle will be inserted into a small cut to remove a sample of the soft tissue inside the bone. Some participants may have a skin biopsy: A small piece of skin will be removed. Some may have a computed tomography (CT) scan: They will lie on a table that slides into a donut-shaped machine that uses X-rays to make pictures of the inside of the body.

Ruxolitinib is a tablet taken by mouth. Participants will take the drug twice a day for up to 6 months.

Participants will have blood tests every week while they are taking the drug. These tests can be done by the participant s own physician and the results sent to the researchers.

Participants will have clinic visits after taking the drug for 3 months and 6 months and then after 1, 2, and 3 years. The blood tests and bone marrow biopsy will be repeated.

Participants who improve while taking the drugs may go on to an extension phase of the study.

DETAILED DESCRIPTION:
Study Description:

This is a prospective, non-randomized, phase I/II study in which participants with relapsed/refractory immune marrow failure (severe aplastic anemia, moderate aplastic anemia, single lineage cytopenias, T-LGL, and hypoplastic MDS) will be treated with the JAK1/2 inhibitor ruxolitinib. Our hypothesis is that JAK1/2 inhibition with ruxolitinib will result in hematologic improvement in participants with immune marrow failure.

Objectives:

The primary objectives are to assess safety and efficacy of the JAK1/2 inhibitor ruxolitinib in immune marrow failure.

The secondary objectives are to assess early and long-term hematologic response, depth of response, development of transfusion independence, rate of relapse, rate of clonal evolution to myeloid malignancy and Paroxysmal Nocturnal Hemoglobinuria (PNH), 3-year overall survival, response after re-initiation of therapy in relapsed participants, maximum tolerated dose.

Endpoints:

The primary endpoints are: (a) the primary safety endpoint will be number of participants who complete a full course of ruxolitinib without cessation required by hematologic toxicity in the 6 months following treatment initiation; (b) The primary efficacy endpoint is overall response (OR) rate by 6 months.

The secondary endpoints are time to OR, OR at 3 months, development of transfusion independence at 3 and 6 months, type of response at 3 and 6 months, rate of relapse up to 3 years, rate of clonal evolution up to 3 years, 3-year overall survival (OS), and number of participants tolerating maximum ruxolitinib dose.

ELIGIBILITY:
* INCLUSION/EXCLUSION CRITERIA:

Participants of both sexes will be considered for inclusion in this study. There will be no racial, ethnic, or sex discrimination. To be eligible to participate in the treatment portion of this study, an individual must meet all of the following inclusion criteria and none of the following exclusion criteria:

INCLUSION CRITERIA:

ALL COHORTS:

* Ability of the participant or legally authorized representative (LAR) to understand and be willing to sign a written informed consent document
* Age 18 or older
* For females of childbearing potential, stated willingness to use an accepted method of contraception for the duration of the study. Accepted methods of contraception are:

  * Total abstinence
  * Use of an implanted or intrauterine hormonal device for at least 30 consecutive days before study drug administration
  * Use of oral, patch or injectable contraceptives or a vaginal hormonal device for at least 30 consecutive days before study drug infusion
  * Use of a non-hormonal intrauterine device for at least 30 consecutive days before study drug administration
  * Two barrier methods such as a diaphragm with spermicide or a condom with spermicide
* For sexually active males with a female partner of childbearing potential, stated willingness to agree to use a condom with spermicide for the duration of the study.
* Diagnosis of immune bone marrow failure (see specific cohort)

COHORT 1: RELAPSED/REFRACTORY SAA:

Meet all 3 criteria below:

Severe aplastic anemia*:

-Bone marrow cellularity <30% excluding lymphocytes

AND

At least two of the following:

* Absolute neutrophil count < 0.5 x 10^9/L
* Platelet count < 20 x 10^9/L
* Absolute Reticulocyte count < 60 x 10^9/L

  * Relapsed or refractory disease as evidenced by a course of at least 1 prior therapy.
  * Not suitable for transplant due to age, co-morbidities, lack of suitable donor, or participant choice.

    * Patients who have a documented historic diagnosis of SAA and have received an ATG-based therapy in the past and are now relapsed / refractory may be included in this cohort even if documentation of original CBC and bone marrow are unavailable.

COHORT 2: RELAPSED/REFRACTORY MODERATE AA:

Moderate AA:

* Aplastic anemia (hypocellular bone marrow for age) with no evidence for other disease processes causing marrow failure, and depression of at least two out of three blood counts below the normal values but not fulfilling the criteria for SAA:

  * Absolute neutrophil count <= l.2 x 10^9/L
  * Platelet count <= 70 x 10^9/L
  * Anemia with hemoglobin <= 9 g/dL and absolute reticulocyte count < 60 x 10^9/L or transfusion dependence
* Relapsed or refractory disease as evidenced by a course of at least 1 prior therapy.

COHORT 3: RELAPSED/REFRACTORY UNILINEAGE BONE MARROW FAILURE DISORDERS:

Cytopenia in lineage as below:

-Erythroid lineage: Hemoglobin <= 9 g/dL and reticulocyte count < 60 x 10^9/L or red cell transfusion dependence and bone marrow with absent or reduced red cell precursors

OR

Platelet lineage: Thrombocytopenia <= 30 x 10^9/L or platelet transfusion dependence and bone marrow with absent or reduced megakaryocytes

OR

Granulocyte lineage: Neutropenia <= 0.5 x 10^9/L and bone marrow for with absent or reduced granulopoiesis

* No evidence of viral or drug suppression of the marrow, T-LGL, dysplasia, or underproduction anemias secondary to B12, folate, iron or other reversible causes.
* Relapsed or refractory disease as evidenced by a course of at least 1 prior therapy.

COHORT 4: RELAPSED/REFRACTORY T-LGL WITH CYTOPENIAS:

* Clinical history supportive of the diagnosis of T-LGL leukemia (i.e., a history of cytopenias with peripheral blood morphologic evidence of LGLs).
* Immunophenotypic studies of peripheral blood showing an increased population of T-LGLs (suggested by staining with CD3+, CD8+ and CD16+ or CD57+) or gamma-delta T cells.
* Restricted or clonal rearrangement of the T-cell receptor by PCR

AND cytopenia as follows:

Severe neutropenia (< 0.5 x 10^9/L);

OR

Severe thrombocytopenia (<= 20 x 10^9/L), or moderate thrombocytopenia (<= 50 x 10^9/L) with active bleeding;

OR

Symptomatic anemia with a hemoglobin <= 9 g/dL or red blood cell transfusion dependence

-Relapsed or refractory disease as evidenced by a course of at least 1 prior therapy.

COHORT 5: HYPOPLASTIC MDS:

-A diagnosis of hypoplastic MDS by WHO 2016, WHO 2022, or ICC criteria with significant cytopenias defined as:

Bone marrow hypocellular for age

AND

Either morphologic dysplasia or cytogenetic abnormality

AND

At least one of the following:

* Neutropenia: Absolute neutrophil count < 0.5 x 10^9/L
* Thrombocytopenia: Platelet count < 30 x 10^9/L or platelet transfusion dependence
* Anemia: Hemoglobin < 9g/dL or red cell transfusion-dependence or absolute reticulocyte count <60 x 10^9/L

  * Relapsed or refractory disease as evidenced by a course of at least 1 prior therapy

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

* Known diagnosis or high suspicion of constitutional marrow failure syndrome
* Evidence of a clonal disorder with poor risk cytogenetics per R-IPSS criteria involving chromosome 7 (-7del/-7), chromosome 3 (inv 3/del3/t(3)) or three or more chromosomal abnormalities (complex)
* MDS with EB-1, EB-2, AML, chronic myelomonocytic leukemia (CMML), MDS/MPN
* For MDS: Has received hypomethylating agent, chemotherapy, or immunomodulatory therapy within 8 weeks prior to study entry
* History of progressive multifocal leuko-encephalopathy (PML)
* Infection not adequately responding to appropriate therapy
* Participants with untreated or poorly controlled HIV, Hepatitis B or C
* Participants with cancer who are on active chemotherapeutic treatment
* Presence of severely impaired renal function defined by CrCl (as calculated by eGFR) less than 15 mL/min not requiring renal dialysis
* Current pregnancy, or unwillingness to take oral contraceptives or use a barrier method of birth control or practice abstinence to refrain from pregnancy if of childbearing potential during this study
* Moribund status or concurrent hepatic, renal, cardiac, neurologic, pulmonary, infectious, or metabolic disease of such severity that it would preclude the participant s ability to tolerate protocol therapy, or that death within 7-10 days is likely
* Inability to understand the investigational nature of the study or to give informed consent or does not have a legally authorized representative or surrogate that can provide informed consent
* Hypersensitivity to ruxolitinib or its components
* Inability to swallow pills
* Currently breastfeeding
* Active non-melanoma skin cancer
* Acute thrombosis (myocardial infarction, ischemic heart disease requiring stents, stroke, pulmonary embolism, or deep venous thrombosis) within the last 6 months
* Patients with a PNH clone >50% who are not taking anticoagulation or anticomplement therapy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Estimated)
Dates: Start 2024-02-20 (Actual); Primary Completion 2030-06-03 (Estimated); Study Completion 2032-06-03 (Estimated)

PRIMARY OUTCOMES:
The number of patients who complete a full course of ruxolitinib without cessation is required by hematologic toxicity. | 6 months
  The primary safety endpoint will be the number of patients who complete a full course of ruxolitinib without cessation required by hematologic toxicity in the 6 months following treatment initiation.
Overall Response Rate. Patients who develop a Complete response at 3 months and stop the drug will also be deemed responders even if they subsequently relapse. | 6 months
  The primary efficacy endpoint is the OR rate by 6 months. Patients who develop CR at 3 months and stop the drug will also be deemed responders even if they subsequently relapse.

SECONDARY OUTCOMES:
Hematological response | 3, 12 months, and yearly thereafter
Depth of response | 3, 6 months
Rate of clonal evolution | Variable
Rate of relapse | Variable
Time to transfusion independence | Variable
Overall survival | Variable
Hematological response of relapse subjects that re-start treatment | Variable
Percent of patients tolerating 20 mg ruxolitinib BID. | Variable

CONTACTS AND LOCATIONS:
Overall Officials: Emma M Groarke, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_001667-H.html